CLINICAL TRIAL: NCT06571084
Title: Establishment and Clinical Application Evaluation of Screening and Diagnostic Cut-off Points With Aldosterone and Renin for Primary Aldosteronism Patients
Brief Title: New Screening and Diagnostic Cut-off Points of PA Patients
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Beijing Anzhen Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Wuhan Asia Heart Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-2260
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Primary Aldosteronism
Keywords: aldosterone; renin; Primary Aldosteronism; cut-off value; diagnosis
MeSH Terms: conditions — Hyperaldosteronism; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All EDTA plasma and some urine samples were stored at -80℃.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- suspected PA: Patients with a high risk for PA who were willing to participate in the study were recruited. The inclusion criteria1 were as follows: persistent hypertension (BP >150/100 mm Hg), or drug-resistant hypertension; newly diagnosed hypertension; hypertension and spontaneous or diuretic-induced hypokalemia; hypertension with adrenal incidentaloma; hypertension and a family history of early-onset hypertension or cerebrovascular accident at a young age (<40 years); or status as a hypertensive first-degree relative of patients with PA; patients with hypertension and obstructive sleep apnea.

SUMMARY:
This study aims to establish the screening and diagnostic cut-off points for primary aldosteronism patients by a novel small molecule "sandwich method" aldosterone and renin chemiluminescent immunoassay.

DETAILED DESCRIPTION:
Primary aldosteronism (PA) is the most common causes of secondary hypertension. The diagnostic workup for PA is composed of multiple steps and requires measurement of both plasma aldosterone and renin. In terms of assay of aldosterone, most of currently available chemiluminescence assays are based on competitive methods. What is actually detected is the sum of aldosterone and its metabolite aldosterone 3C glucuronide, which causes the value to be about 50%~100% higher than the actual value. This study aims to establish a new ARR (aldosterone/renin ratio) cutoff point for PA screening and a new cutoff point for PA diagnosis, using a recently developed two-site sandwich chemiluminescence method (Snibe, China) for aldosterone and renin assay.

Hypertensive patients referred to hospitals for screening of PA will be included. All the participants proceed to seated saline infusion test (SIT) and captopril challenge test (CCT) for confirmation. Aldosterone and renin will be measured using chemiluminescent immunoassay on the Liaison analyzer (DiaSorin, Italy) and MAGLUMI X8 (Snibe, China), as well as liquid chromatography-tandem mass spectrometry (LC-MS/MS) platform. According to the experience of Fuwai Hospital, the following diagnosis criteria are proposed: Based on the results of currently used (DiaSorin, Italy), aldosterone > 8.5ng/dL and renin < 15μIU/mL after sitting saline infusion conform PA, and aldosterone ≤ 8.5ng/dL excludes PA.

The total number of cases to be enrolled in this study is planned to be 770, including at least 77 positive subjects and at least 406 negative subjects. By drawing the ROC curve, the point corresponding to the maximum value of the Youden index will be selected as the cutoff value, and the corresponding sensitivity, specificity, positive predictive value, negative predictive value, positive likelihood ratio, negative likelihood ratio, etc. will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* 18-75y;
* persistent hypertension (BP >150/100 mm Hg), or drug-resistant hypertension;
* newly diagnosed hypertension;
* hypertension and spontaneous or diuretic-induced hypokalemia;
* hypertension with adrenal incidentaloma;
* hypertension and a family history of early-onset hypertension or cerebrovascular accident at a young age (<40 years);
* status as a hypertensive first-degree relative of patients with PA;
* patients with hypertension and obstructive sleep apnea.

Exclusion Criteria:

* age <18; BMI ≤ 18.0kg/m2 or ≥ 35.0 kg/m2;
* a diagnosis of secondary hypertension other than PA;
* chronic cardiac dysfunction (NYHA III-IV);
* medium and several kidney dysfunction (Ccr<30ml/min);
* liver cirrhosis;
* terminal malignant tumor;
* recent use of steroids or oral contraceptives;
* pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-75 years old and highly suspected primary aldosteronism will be included. Patients will be excluded if who is secondary hypertension other than PA, chronic cardiac dysfunction (NYHA III-IV), medium and several kidney dysfunction (Ccr<30ml/min), with history of liver cirrhosis, oncosis and recent use of steroids or oral contraceptives, pregnant or lactating.
Sampling Method: Non-Probability Sample
Enrollment: 770 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Preliminary confirmation positive for primary aldosteronism | 1 month
  Aldosterone ≥ 85pg/ml after sitting saline test

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cai, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital; Zhou Zhou, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Kai-juan Wang, Beijing, China

IPD SHARING:
Plan to Share IPD: No